CLINICAL TRIAL: NCT02579759
Title: International, Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Study Assessing in Parallel Groups the Efficacy and Safety of 2 Doses of PXT3003 in Patients With Charcot-Marie-Tooth Disease Type 1A Treated 15 Months
Brief Title: Phase III Trial Assessing the Efficacy and Safety of PXT3003 in CMT1A Patients (PLEO-CMT)
Acronym: PLEO-CMT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharnext S.C.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLN-PXT3003-02; 2015-002378-19 (EudraCT Number)
Record Dates: First submitted 2015-09-28; First posted 2015-10-20 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Charcot-Marie-Tooth Disease Type 1A
Keywords: PXT3003
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PXT3003 dose 1 (Active Comparator): Oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months
  Interventions: Drug: PXT3003 dose 1
- PXT3003 dose 2 (Active Comparator): Oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months
  Interventions: Drug: PXT3003 dose 2
- placebo (Placebo Comparator): Oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PXT3003 dose 1 — Liquid oral solution, 5 ml twice a day, morning and evening with food
  Other Names: DOSE 1
  Arms: PXT3003 dose 1
Drug: PXT3003 dose 2 — Liquid oral solution, 5 ml twice a day, morning and evening with food
  Other Names: DOSE 2
  Arms: PXT3003 dose 2
Drug: placebo — Liquid oral solution, 5 ml twice a day, morning and evening with food
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether PXT3003 is effective and safe in the treatment of Charcot-Marie-Tooth disease - Type 1 A (CMT1A). This double-blind study will assess in parallel groups 2 doses of PXT3003 compared to Placebo in CMT1A patients treated for 15 months.

DETAILED DESCRIPTION:
PXT3003 is a fixed dose combination of (RS)-baclofen, naltrexone hydrochloride and D-sorbitol selected via a Systems Biology approach and developed by Pharnext, with the aim to limit the production of PMP22 and protect/improve axonal function in patients with CMT1A. On September 18th 2017, PXT3003 dose 2 was prematurely discontinued, due to an unexpected investigational medicinal product quality event (failed month 18 stability testing). This resulted in a large proportion of missing data that led us to reconsider the efficacy analysis that was initially planned in the protocol.The independent data safety monitoring committee did not identify any safety concern on September 5th 2017. All patients randomised to dose 2 were requested to undergo the end of study visit, and were offered to enter the extension study (CLN-PXT3003-03).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 16 to 65 years;
* Patient with a proven genetic diagnosis of CMT1A;
* Mild-to-moderate severity assessed by Charcot-Marie-Tooth Neuropathy Score (version 2) with a score >2 and ≤18;
* Muscle weakness in at least foot dorsiflexion;
* Motor nerve conduction of the ulnar nerve of at least 15 m/sec;
* Providing signed written informed consent to participate in the study and willing and able to comply with all study procedures and scheduled visits.

Exclusion Criteria:

* Any other associated cause of peripheral neuropathy such as diabetes;
* Patient with another significant neurological disease or a concomitant major systemic disease;
* Clinically significant history of unstable medical illness since the last 30 days (unstable angina, cancer…) that may jeopardize the participation in the study;
* Significant hematologic disease, hepatitis or liver failure, renal failure;
* Limb surgery within six months before randomization or planned before trial completion;
* Clinically significant abnormalities on the pre-study laboratory evaluation, physical evaluation, electrocardiogram (ECG);
* Elevated ASAT/ALAT (> 3 x ULN) and elevated serum creatinine levels (> 1.25 x ULN);
* History of recent alcohol or drug abuse or non-adherence with treatment or other experimental protocols;
* Patient using unauthorized concomitant treatments including but not limited to baclofen, naltrexone, sorbitol (pharmaceutical form), opioids, levothyroxin and potentially neurotoxic drugs such as amiodarone, chloroquine, cancer drugs susceptible to induce a peripheral neuropathy. Patient who can/agrees to stop these medications 4 weeks before randomization and during the whole study duration can be included;
* Female of childbearing potential (apart of patient using adequate contraceptive measures), pregnant or breast feeding;
* Known hypersensitivity to any of the individual components of PXT3003;
* Porphyria as it is a contra indication to baclofen, and it may also induce neuropathy;
* Suspected inability to complete the study follow-up (foreign workers, transient visitors, tourists or any others for whom follow-up evaluation is not assured);
* Limited mental capacity or psychiatric disease rendering the subject unable to provide written informed consent or comply with evaluation procedures;
* Patient who has participated in another trial of investigational drug(s) within the past 30 days;
* If a patient from the same family, living in the same household, has already been included in this study, it will not be possible to include another patient from the same family to avoid mixing of therapeutic units; therefore there would be a risk of inversion of the blind treatments which could jeopardize the interpretation of study results.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahram Attarian, MD, Principal Investigator — CHU La Timone, Marseille, France; Peter Young, MD, Principal Investigator — University Hospital Munster, Germany; Teresa Sevilla, MD, Principal Investigator — Hospital Universitari i Politécnic La Fe, Valencia, Spain; Marianne De Visser, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Philip Van Damme, MD, Principal Investigator — UZ Leuven, Belgium; Mark Roberts, MD, Principal Investigator — Salford Royal NHS Foundation Trust, Manchester, UK; Florian Thomas, MD, Principal Investigator — Saint-Louis University, Saint-Louis, USA; Jack Puymirat, MD, Principal Investigator — University Hospital of Quebec
Locations (30):
- United States (11):
  - Department of Neurology, Cedars-Sinai Medical Center, Los Angeles, California
  - Hospital for Special Care, New Britain, New Britain, Connecticut
  - Department of Neurology, McKnight Brain Institute, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Department of Neurology, University of Minnesota, Minneapolis, Minnesota
  - Department of Neurology and Psichiatry, Saint Louis University, St Louis, Missouri
  - Peripheral Neuropathy Center, Neurological Institue Building, Columbia University Medical Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Saint Luke's Rehabilitation Institute, Spokane, Washington
- Departement of Neurology, UZ Leuven, Leuven, Belgium
- University Hospital of Quebec, Québec, Quebec, Canada
- France (6):
  - Centre de Référence des Maladies Neuromusculaires, Hôpital Swynghedauwl, CHU de Lille, Lille
  - Centre de Référence des Neuropathies Périphériques Rares, Hôpital Dupuytren, CHU Limoges, Limoges
  - Service de Neurologie et du Sommeil, CHU Lyon Sud, Lyon
  - Centre de Référence des Maladies Neuromusculaires, Pôle des Neurosciences Clinique, CHU la Timone, Marseille
  - Centre de Référence des Maladies Neuromusculaires; Hôtel Dieu, CHU de Nantes, Nantes
  - Service de Neurologie, Hôpital Kremlin Bicêtre, Paris
- Germany (4):
  - Department of Neurology and Institute for Neuropathology, University Hospital RWTH Aachen, Aachen
  - Department of Clinical Neurophysiology, University Medical Center Göttingen, Göttingen
  - Department of Neurology, Ludwig-Maximillian University, Munich, Munich
  - Department for Sleep Medicine and Neuromuscular, University Hospital Münster, Münster
- Departement of Neurology, Academic Medical Center, Amsterdam, Netherlands
- Spain (4):
  - Department of neurology, Hospital Univesitario de Bellvitge, Barcelona
  - Servicio de Neurologia, Hospital Universitario La Paz, Madrid
  - Centro de Diagnostico y Tratamiento, Hospital Universitario Virgen del Rocio, Seville
  - Servicio de Neurologia, Hospital Univesitari i Politécnic La Fe, Valencia
- United Kingdom (2):
  - Department of Neurology, Salford Royal NHS Foundation Trust, Salford, Manchester
  - Ninewells Hospital and Medical School, Dundee, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Attarian S, Vallat JM, Magy L, Funalot B, Gonnaud PM, Lacour A, Pereon Y, Dubourg O, Pouget J, Micallef J, Franques J, Lefebvre MN, Ghorab K, Al-Moussawi M, Tiffreau V, Preudhomme M, Magot A, Leclair-Visonneau L, Stojkovic T, Bossi L, Lehert P, Gilbert W, Bertrand V, Mandel J, Milet A, Hajj R, Boudiaf L, Scart-Gres C, Nabirotchkin S, Guedj M, Chumakov I, Cohen D. An exploratory randomised double-blind and placebo-controlled phase 2 study of a combination of baclofen, naltrexone and sorbitol (PXT3003) in patients with Charcot-Marie-Tooth disease type 1A. Orphanet J Rare Dis. 2014 Dec 18;9:199. doi: 10.1186/s13023-014-0199-0. PMID 25519680
- [Result] Chumakov I, Milet A, Cholet N, Primas G, Boucard A, Pereira Y, Graudens E, Mandel J, Laffaire J, Foucquier J, Glibert F, Bertrand V, Nave KA, Sereda MW, Vial E, Guedj M, Hajj R, Nabirotchkin S, Cohen D. Polytherapy with a combination of three repurposed drugs (PXT3003) down-regulates Pmp22 over-expression and improves myelination, axonal and functional parameters in models of CMT1A neuropathy. Orphanet J Rare Dis. 2014 Dec 10;9:201. doi: 10.1186/s13023-014-0201-x. PMID 25491744
- [Result] Mandel J, Bertrand V, Lehert P, Attarian S, Magy L, Micallef J, Chumakov I, Scart-Gres C, Guedj M, Cohen D. A meta-analysis of randomized double-blind clinical trials in CMT1A to assess the change from baseline in CMTNS and ONLS scales after one year of treatment. Orphanet J Rare Dis. 2015 Jun 13;10:74. doi: 10.1186/s13023-015-0293-y. PMID 26070802
- [Result] Prukop T, Stenzel J, Wernick S, Kungl T, Mroczek M, Adam J, Ewers D, Nabirotchkin S, Nave KA, Hajj R, Cohen D, Sereda MW. Early short-term PXT3003 combinational therapy delays disease onset in a transgenic rat model of Charcot-Marie-Tooth disease 1A (CMT1A). PLoS One. 2019 Jan 16;14(1):e0209752. doi: 10.1371/journal.pone.0209752. eCollection 2019. PMID 30650121
- [Result] Hajj R, Prukop T, Wernick S, Ewers D, Brureau A, Cholet N, Laffaire J, Nave KA, Cohen D, Sereda M. Baclofen, Naltrexone and Sorbitol all contribute to the efficacy of PXT3003 in CMT1A Rats. EMJ Neurol, 2019;7[1]:47-49
- [Result] Attarian S, Vallat JM, Magy L, Funalot B, Gonnaud PM, Lacour A, Pereon Y, Dubourg O, Pouget J, Micallef J, Franques J, Lefebvre MN, Ghorab K, Al-Moussawi M, Tiffreau V, Preudhomme M, Magot A, Leclair-Visonneau L, Stojkovic T, Bossi L, Lehert P, Gilbert W, Bertrand V, Mandel J, Milet A, Hajj R, Boudiaf L, Scart-Gres C, Nabirotchkin S, Guedj M, Chumakov I, Cohen D. Erratum to: An exploratory randomised double-blind and placebo-controlled phase 2 study of a combination of baclofen, naltrexone and sorbitol (PXT3003) in patients with Charcot-Marie-Tooth disease type 1A. Orphanet J Rare Dis. 2016 Jul 7;11(1):92. doi: 10.1186/s13023-016-0463-6. No abstract available. PMID 27387831
- See also: Attarian et al., 2016 — https://www.ncbi.nlm.nih.gov/pubmed/25519680
- See also: Chumakov et al., 2014 — https://www.ncbi.nlm.nih.gov/pubmed/?term=25491744
- See also: Mandel et al., 2015 — https://www.ncbi.nlm.nih.gov/pubmed/?term=26070802
- See also: Prukop et al., 2019 — https://www.ncbi.nlm.nih.gov/pubmed/?term=30650121
- See also: Attarian et al., Erratum, 2016 — https://www.ncbi.nlm.nih.gov/pubmed/?term=27387831
- See also: Hajj et al., 2019 — https://www.emjreviews.com/neurology/abstract/baclofen-naltrexone-and-sorbitol-all-contribute-to-the-efficacy-of-pxt3003-in-cmt1a-rats/

RESULTS

PARTICIPANT FLOW:
Groups:
- PXT3003 Dose 1: Liquid oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months.
  PXT3003 dose 1: 3 mg baclofen, 0.35 mg naltrexone and 105 mg sorbitol (twice a day, morning and evening with food).
- PXT3003 Dose 2: Liquid oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months.
  PXT3003 dose 2: 6 mg baclofen, 0.70 mg naltrexone and 210 sorbitol (twice a day, morning and evening with food).
- Placebo: Liquid oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months.
  PXT3003 matching placebo had the same presentation, the same aspect and taste in order to be undistinguishable (twice a day, morning and evening with food).
Period: Overall Study
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Started | 109 | 113 | 101
Completed (Completed at 12 months) | 85 | 49 | 80
Not Completed | 24 | 64 | 21
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Other (Sponsor stopped Dose 2) | 0 | 1 | 0
Not completed — BfArM hold | 13 | 12 | 12
Not completed — Sponsor stopped Dose 2 | 0 | 41 | 0
Not completed — Non compliance | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Inclusion/exclusion criteria | 0 | 0 | 1
Not completed — Adverse Event | 4 | 3 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 5
Not completed — Lost to Follow-up | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo | Total
Number analyzed (Participants) | 109 | 113 | 101 | 323
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 8 | 2 | 15
  Between 18 and 65 years | 103 | 104 | 97 | 304
  >=65 years | 1 | 1 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.3) | 39.6 (13.9) | 42.1 (13.2) | 40.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 68 | 62 | 190
  Male | 49 | 45 | 39 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 108 | 111 | 100 | 319
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 4 | 5 | 14
  Netherlands | 2 | 3 | 3 | 8
  Belgium | 4 | 6 | 5 | 15
  United States | 21 | 24 | 18 | 63
  United Kingdom | 2 | 0 | 1 | 3
  France | 31 | 31 | 29 | 91
  Germany | 22 | 23 | 22 | 67
  Spain | 22 | 22 | 18 | 62

OUTCOME MEASURES:

1. Primary Outcome: Overall Neuropathy Limitation Scale (ONLS) Total Score
Description: The primary efficacy variable used in the main analysis is the mean of the available ONLS values at month 12 and month 15.
  The ONLS is a disability scale that was derived and improved from the Overall Disability Sum Score (ODSS) to measure limitations in the everyday activities of the upper limbs (rated on 5 points) and the lower limbs (rated on 7 points). The total score is a 12-point scale: 0 (no disability) to 12 (maximum disability). Lower values in the ONLS indicate a better clinical condition.
  Reported values are the values at Baseline (Base) and the average of the available values at Month 12 and Month 15 (Fin).
Time Frame: From Baseline to Month 15
Population: mFAS selection
Measure: Mean (Standard Deviation); unit: Scores on the ONLS
Groups:
- Placebo: Oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months.
  PXT3003 matching placebo had the same presentation, the same aspect and taste in order to be undistinguishable (twice a day, morning and evening with food).
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 93 | 55 | 87
Scores on the ONLS
  Base | 3.33 (1.05) | 3.05 (1.13) | 3.23 (1.19)
  Fin | 3.25 (1.00) | 2.82 (1.28) | 3.36 (1.16)
Statistical Analysis 1: Comparison: PXT3003 Dose 2 vs Placebo; The main analysis was performed as follows: 1. Analysis population: modified Full Analysis Set (mFAS) 2. Statistical model: ANCOVA where the mean at 12 and 15 months of each treatment group was compared against the placebo group, adjusting for the baseline value and assuming centre as a random effect 3. Missing value imputation: multiple imputation taking into account the reason of missingness; Test type: Superiority; p = 0.008, ANCOVA; Mean Difference (Final Values) = -0.37, 97.5% CI 2-sided [-0.68 to -0.06], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: PXT3003 Dose 1 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.287, ANCOVA; Mean Difference (Final Values) = -0.13, 97.5% CI 2-sided [-0.39 to 0.14], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: PXT3003 Dose 2 vs Placebo; This analysis was performed as follows: 1. Analysis population: modified Full Analysis Set (mFAS) 2. Statistical model: Longitudinal model where the effect of each treatment over time (baseline, 6, 12 and 15 months) was estimated through a mixed model with repeated measures (MMRM) assuming time from baseline (Time) and Time-by-Treatment full interaction as fixed effects and patient as random effect and considering Time as continuous linear effect 3. Missing value imputation: No imputation; Test type: Superiority; p = 0.013, Longitudinal mixed model; Mean Difference (Final Values) = -0.31, 97.5% CI 2-sided [-0.59 to -0.03], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: PXT3003 Dose 1 vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.05, Longitudinal mixed model; Mean Difference (Final Values) = -0.19, 97.5% CI 2-sided [-0.42 to 0.03], Standard Error of Mean 0.1
Statistical Analysis 5: Comparison: PXT3003 Dose 1 vs PXT3003 Dose 2 vs Placebo; Dose effect: Dose is defined as a numerical variable proportional to quantity of PXT3003 administered (0 for Placebo, 1 for Dose 1, 2 for Dose 2). The analysis was performed as follows: 1. Analysis population: modified Full Analysis Set (mFAS) 2. Statistical model: ANCOVA assessing the dose-effect at the mean of 12 and 15 months, adjusting for baseline value and assuming centre as random effect 3. Missing value imputation: multiple imputation taking into account the reason of missingness; Test type: Superiority; p = 0.013, Regression, Linear; Slope = -0.17, 95% CI 2-sided [-0.31 to -0.04], Standard Error of Mean 0.07

2. Secondary Outcome: Mean of Ten Meter Walking Test (10MWT)
Description: This outcome measure is the mean of the available 10MWT values at month 12 and month 15.
  The 10MWT is a simple to administer, standardized, reliable and valid evaluation of functional exercise capacity and gait that has been used to evaluate neurologic disorders and CMT patients.
  Lower Time to Walk 10 Meters values indicate a better clinical condition.
  Reported values are the values at Baseline (Base) and the average of the available values at Month 12 and Month 15 (Fin).
Time Frame: From Baseline to Month 15
Population: mFAS selection
Measure: Mean (Standard Deviation); unit: Seconds (s)
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 93 | 55 | 87
Seconds (s)
  Base | 6.93 (1.77) | 7.14 (1.77) | 7.28 (1.91)
  Fin | 6.47 (1.59) | 6.52 (1.39) | 6.91 (1.82)
Statistical Analysis 1: Comparison: PXT3003 Dose 2 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.016, ANCOVA; Mean Difference (Final Values) = -0.47, 97.5% CI 2-sided [-0.91 to -0.03], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: PXT3003 Dose 1 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.084, ANCOVA; Mean Difference (Final Values) = -0.28, 97.5% CI 2-sided [-0.65 to 0.08], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: PXT3003 Dose 1 vs PXT3003 Dose 2 vs Placebo; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.015, Regression, Linear; Slope = -0.22, 95% CI 2-sided [-0.41 to -0.04], Standard Error of Mean 0.09

3. Secondary Outcome: Mean of the CMTNS-v2 Sensory Score
Description: This outcome measure is the mean of the available CMTNS-v2 Sensory Score values at month 12 and month 15.
  The CMTNS-v2 is a specific scale designed to assess severity of impairment in CMT disease. It is a 36-point scale based on nine items to quantify impairment (sensory symptoms, pin sensibility, vibration and arm and leg strength), activity limitations (motor symptoms arms and legs) and electrophysiological function (amplitudes of ulnar CMAP and SNAP). The CMTNS-v2 goes from 0 (no impairment) to 36 (maximum impairment) whom each sub-items goes from 0 to 4.
  The CMTNS-v2 Sensory score is summed of items 1+4+5 of CMTNS-v2 (Sensory symptoms, Pinprick sensibility and Vibration). It is a 12-point score: 0 (no impairment) to 12 (maximum impairment).
  Lower CMTNS-v2 Sensory Score values indicate a better clinical condition.
  Reported values are the values at Baseline (Base) and the average of the available values at Month 12 and Month 15 (Fin).
Time Frame: From Baseline to Month 15
Population: mFAS selection
Measure: Mean (Standard Deviation); unit: Scores on the CMTNS-v2 Sensory Score
Groups:
- Placebo: Oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months
  PXT3003 matching placebo had the same presentation, the same aspect and taste in order to be undistinguishable (twice a day, morning and evening with food).
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 93 | 55 | 87
Scores on the CMTNS-v2 Sensory Score
  Base | 5.00 (2.28) | 4.47 (2.21) | 4.97 (2.04)
  Fin | 4.55 (1.96) | 4.23 (2.38) | 4.68 (2.14)
Statistical Analysis 1: Comparison: PXT3003 Dose 2 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.162, ANCOVA; Mean Difference (Final Values) = -0.39, 97.5% CI 2-sided [-1.01 to 0.23], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: PXT3003 Dose 1 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.556, ANCOVA; Mean Difference (Final Values) = -0.14, 97.5% CI 2-sided [-0.66 to 0.39], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: PXT3003 Dose 1 vs PXT3003 Dose 2 vs Placebo; Dose is defined as a numerical variable proportional to quantity of PXT3003 administered (0 for Placebo, 1 for Dose 1, 2 for Dose 2). The analysis was performed as follows: 1. Analysis population: modified Full Analysis Set (mFAS) 2. Statistical model: ANCOVA assessing the dose-effect at the mean of 12 and 15 months, adjusting for baseline value and assuming centre as random effect 3. Missing value imputation: multiple imputation taking into account the reason of missingness; Test type: Superiority; p = 0.204, Regression, Linear; Slope = -0.17, 95% CI 2-sided [-0.43 to 0.09], Standard Error of Mean 0.13

4. Secondary Outcome: Mean of the CMTNS-v2 Examination Score (CMTES-v2)
Description: This outcome measure is the mean of the available CMTNS-v2 Examination Score values at month 12 and month 15.
  The CMTNS-v2 is a specific scale designed to assess severity of impairment in CMT disease. It is a 36-point scale based on nine items to quantify impairment (sensory symptoms, pin sensibility, vibration and arm and leg strength), activity limitations (motor symptoms arms and legs) and electrophysiological function (amplitudes of ulnar CMAP and SNAP). The CMTNS-v2 goes from 0 (no impairment) to 36 (maximum impairment) whom each sub-items goes from 0 to 4.
  The CMTES-v2 is summed of item 1 to 7 of the CMTNS-v2 (limited to impairment items and excluding electrophysiological items). It is a 28-point score: 0 (no impairment) to 28 (maximum impairment).
  Lower CMTES-v2 values indicate a better clinical condition.
  Reported values are the values at Baseline (Base) and the average of the available values at Month 12 and Month 15 (Fin).
Time Frame: From Baseline to Month 15
Population: mFAS selection
Measure: Mean (Standard Deviation); unit: Scores on the CMTES-v2
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 93 | 55 | 87
Scores on the CMTES-v2
  Base | 9.49 (2.80) | 8.78 (2.73) | 9.51 (2.79)
  Fin | 9.01 (2.62) | 8.24 (3.13) | 9.02 (3.05)
Statistical Analysis 1: Comparison: PXT3003 Dose 2 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.232, ANCOVA; Mean Difference (Final Values) = -0.43, 97.5% CI 2-sided [-1.25 to 0.38], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: PXT3003 Dose 1 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.868, ANCOVA; Mean Difference (Final Values) = -0.05, 97.5% CI 2-sided [-0.74 to 0.64], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: PXT3003 Dose 1 vs PXT3003 Dose 2 vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.322, Regression, Linear; Slope = -0.18, 95% CI 2-sided [-0.53 to 0.17], Standard Error of Mean 0.18

5. Secondary Outcome: Mean of the Results at the Nine-Hole Peg Test (9-HPT)
Description: This outcome measure is the mean of the available 9-HPT values at month 12 and month 15.
  The Nine-Hole Peg Test (9HPT) is a simple timed test of fine motor coordination of extremitied in the upper limbs. It measures the time needed by the patient to insert 9 pegs in nine holes and to remove them (normal required time 18 seconds).
  Lower 9HPT values indicate a better clinical condition.
  Reported values are the values at Baseline (Base) and the average of the available values at Month 12 and Month 15 (Fin).
Time Frame: From Baseline to Month 15
Population: mFAS selection
Measure: Mean (Standard Deviation); unit: Seconds (s)
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 93 | 55 | 87
Seconds (s)
  Base | 25.62 (5.60) | 27.33 (11.15) | 25.18 (4.41)
  Fin | 23.85 (4.52) | 25.67 (8.29) | 24.41 (4.01)
Statistical Analysis 1: Comparison: PXT3003 Dose 2 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.377, ANCOVA; Mean Difference (Final Values) = -0.4, 97.5% CI 2-sided [-1.43 to 0.62], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: PXT3003 Dose 1 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.334, ANCOVA; Mean Difference (Final Values) = -0.36, 97.5% CI 2-sided [-1.21 to 0.48], Standard Error of Mean 0.38
Statistical Analysis 3: Comparison: PXT3003 Dose 1 vs PXT3003 Dose 2 vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.373, Regression, Linear; Slope = -0.19, 95% CI 2-sided [-0.62 to 0.23], Standard Error of Mean 0.22

6. Secondary Outcome: Number of Subjects With at Least One TEAE
Description: Safety selection was to include all randomized patients that have received at least one dose of study treatment.
  Safety and tolerability of PXT3003 were compared to placebo on the incidence of treatment-emergent adverse events (TEAEs); they were evaluated by type/nature, severity/intensity, seriousness, and relationship to study drug.
Time Frame: The period between the patient signing the informed consent and 30 days after the end of study (i.e. completion/early discontinuation/last contact as recorded on the 'Study Completion on Early Termination' form up to 15 months)
Population: FAS selection
Measure: Number; unit: participants
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 109 | 113 | 101
participants
  Any TEAE | 89 | 87 | 83
  Any related TEAE | 39 | 38 | 34
  Any moderately severe or severe related TEAE | 8 | 5 | 10

7. Secondary Outcome: Incidence of AE Leading to Withdrawal of Study Drug
Description: Safety and tolerability of PXT3003 were compared to placebo on the incidence of TEAEs leading to withdrawal of study drug.
Time Frame: as for outcome 6
Population: FAS selection
Measure: Number; unit: participants
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 109 | 113 | 101
participants
  Any TEAE leading to drug withdrawal | 6 | 6 | 6
  Any related TEAE leading to drug withdrawal | 3 | 2 | 2

8. Secondary Outcome: Incidence of SAEs
Description: Safety and tolerability of PXT3003 were compared to placebo on the incidence of serious adverse events (SAEs).
Time Frame: as for outcome 6
Population: FAS selection
Measure: Number; unit: participants
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 109 | 113 | 101
participants
  Any serious TEAE | 10 | 3 | 5
  Any related serious TEAE | 0 | 0 | 0
  Any serious TEAE leading to drug withdrawal | 1 | 0 | 0

9. Other Pre Specified Outcome: Mean of the CMTNS-v2 Sensory Symptoms
Description: This outcome measure is the mean of the available CMTNS-v2 Sensory Symptoms values at month 12 and month 15.
  The CMTNS-v2 is a specific scale designed to assess severity of impairment in CMT disease. It is a 36-point scale based on nine items to quantify impairment (sensory symptoms, pin sensibility, vibration and arm and leg strength), activity limitations (motor symptoms arms and legs) and electrophysiological function (amplitudes of ulnar CMAP and SNAP). The CMTNS-v2 goes from 0 (no impairment) to 36 (maximum impairment) whom each sub-items goes from 0 to 4.
  The CMTNS-v2 Sensory Symptoms is the first item of the CMTNS-v2. It is a 4-point score: 0 (no impairment) to 4 (maximum impairment).
  Lower CMTNS-v2 Sensory Symptoms values indicate a better clinical condition.
  Reported values are the values at Baseline (Base) and the average of the available values at Month 12 and Month 15 (Fin).
Time Frame: From Baseline to Month 15
Population: mFAS selection
Measure: Mean (Standard Deviation); unit: Scores on the CMTNS-v2 Sensory Symptoms
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 93 | 55 | 87
Scores on the CMTNS-v2 Sensory Symptoms
  Base | 1.26 (0.95) | 0.96 (0.98) | 1.09 (0.90)
  Fin | 1.18 (0.81) | 0.93 (0.96) | 1.21 (0.94)
Statistical Analysis 1: Comparison: PXT3003 Dose 2 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.023, ANCOVA; Mean Difference (Final Values) = -0.29, 97.5% CI 2-sided [-0.58 to 0], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: PXT3003 Dose 1 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.162, ANCOVA; Mean Difference (Final Values) = -0.15, 97.5% CI 2-sided [-0.4 to 0.09], Standard Error of Mean 0.11

10. Other Pre Specified Outcome: Plasma Concentrations of Baclofen at Trough and at 90 Min After Drug Intake
Description: Plasma concentration of PXT3003 components were measured at trough (prior to dose) and 90 minutes after drug intake.
  The mean plasma values of the baseline correspond to half of the administered dose.
Time Frame: At Month 12 and Month 15
Population: PP selection LLOQ = 30 pg/mL The placebo arm has not been described for this endpoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2
Number analyzed (Participants) | 68 | 38
pg/mL
  At trough, at Month 12 | 13739.3 (20313.6) | 11651.9 (6151.1)
  At trough, at Month 15 | 9009.7 (10910.3) | 8686.6 (9172.8)
  At 90 min after drug intake, at Month 12 | 52201.6 (21494.6) | 90238.7 (29972.8)
  At 90 min after drug intake, at Month 15 | 47021.1 (19834.5) | 105825.4 (38756.7)

11. Other Pre Specified Outcome: Plasma Concentrations of Naltrexone at Trough and at 90 Min After Drug Intake
Description: as for outcome 10
Time Frame: At Month 12 and month 15
Population: PP selection LLOQ = 30 pg/mL The placebo arm has not been described for this endpoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2
Number analyzed (Participants) | 68 | 38
pg/mL
  At trough, at Month 12 | 33.0 (15.8) | 42.0 (66.0)
  At trough, at Month 15 | 31.8 (14.0) | 30.0 (0.0)
  At 90 min after drug intake, at Month 12 | 63.0 (47.4) | 107.5 (88.6)
  At 90 min after drug intake, at Month 15 | 55.0 (39.3) | 130.9 (81.4)

12. Other Pre Specified Outcome: Plasma Concentrations of 6β-naltrexol at Trough and at 90 Min After Drug Intake
Description: Plasma concentration of PXT3003 components were measured at trough (prior to dose) and peak (90 minutes post dose).
  The mean plasma values of the baseline correspond to half of the administered dose.
Time Frame: At Month 12 and Month 15
Population: PP selection LLOQ = 50 pg/mL The placebo arm has not been described for this endpoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2
Number analyzed (Participants) | 68 | 38
pg/mL
  At trough, at Month 12 | 290.1 (177.4) | 526.4 (245.6)
  At trough, at Month 15 | 260.4 (121.8) | 352.3 (319.0)
  At 90 min after drug intake, at Month 12 | 632.5 (230.1) | 1257.1 (454.3)
  At 90 min after drug intake, at Month 15 | 586.4 (205.4) | 1450.9 (438.0)

13. Other Pre Specified Outcome: Number of Participants With ONLS Therapy Response 1
Description: ONLS Therapy Response 1 was defined as the number of participants (responders) with an improvement on final ONLS Total Score of at least one point. A higher response rate indicate a better clinical condition.
Time Frame: From Baseline to Month 15
Population: Completers selection
Measure: Number; unit: Number of Participants
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 85 | 49 | 80
Number of Participants | 16 | 14 | 14
Statistical Analysis 1: Comparison: PXT3003 Dose 2 vs Placebo; The proportion of responders (on Completers selection only) at the end of treatment was assessed through a Generalized Linear Mixed Model (GLMM) featuring logistic regression including treatment as a fixed effect, adjusting for the baseline value and center as a random effect; Test type: Superiority; p = 0.097, General Linear Mixed Model; Odds Ratio (OR) = 2.09, 97.5% CI 2-sided [0.77 to 5.68]
Statistical Analysis 2: Comparison: PXT3003 Dose 1 vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.865, General Linear Mixed Model; Odds Ratio (OR) = 1.07, 97.5% CI 2-sided [0.42 to 2.7]

14. Other Pre Specified Outcome: Number of Participants With ONLS Therapy Response 2
Description: ONLS Therapy Response 2 was defined as the number of participants with no deterioration (responders) on final ONLS Total Score.
  A higher response rate indicates a better clinical condition.
Time Frame: From Baseline to Month 15
Population: Completers selection
Measure: Number; unit: Number of Participants
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
Number analyzed (Participants) | 85 | 89 | 80
Number of Participants | 66 | 42 | 58
Statistical Analysis 1: Comparison: PXT3003 Dose 2 vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.026, General Linear Mixed Model; Odds Ratio (OR) = 3.39, 97.5% CI 2-sided [0.99 to 11.62]
Statistical Analysis 2: Comparison: PXT3003 Dose 1 vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.569, General Linear Mixed Model; Odds Ratio (OR) = 1.26, 97.5% CI 2-sided [0.5 to 3.16]

ADVERSE EVENTS:
Time Frame: The AE reporting period therefore started with the subject signing the informed consent form and ended 30 days after the end of study (corresponding to the date of "Date of completion/early discontinuation/last contact" recorded in the termination module up to 15 months)
Description: This definition was extended due to the discontinuation of Dose 2 and study on hold in Germany. The period of AE reporting was extended to 1 month after the end of study, without informed consent signed for study CLN-PXT3003-03 during this period.
  Only Treatment-Emergent Adverse Events (TEAE) have been reported for non-serious advers events.
Groups:
- PXT3003 Dose 1: Oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months.
  PXT3003 dose 1: 3 mg baclofen, 0.35 mg naltrexone and 105 mg sorbitol (twice a day, morning and evening with food).
- PXT3003 Dose 2: Oral solution, 5 ml b.i.d. (taken morning and evening with food) during 15 months.
  PXT3003 dose 2: 6 mg baclofen, 0.70 mg naltrexone and 210 sorbitol (twice a day, morning and evening with food).
Arm/Group | PXT3003 Dose 1 | PXT3003 Dose 2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/113 | 0/101
Serious Adverse Events (participants affected / at risk) | 10/109 | 3/113 | 5/101
Other Adverse Events (participants affected / at risk) | 89/109 | 87/113 | 83/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PXT3003 Dose 1 (N=109) | PXT3003 Dose 2 (N=113) | Placebo (N=101)
Arthrolysis (Surgical and medical procedures) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Median nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Congenital foot malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PXT3003 Dose 1 (N=109) | PXT3003 Dose 2 (N=113) | Placebo (N=101)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Asthenia (General disorders) | 3 (3) | 2 (2) | 7 (9) — and administation site conditions
Fatigue (General disorders) | 11 (15) | 2 (2) | 6 (6) — and administation site conditions
Influenza like illness (General disorders) | 3 (5) | 6 (9) | 0 (0) — and administation site conditions
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 2 (2) — and administation site conditions
Anxiety (Psychiatric disorders) | 3 (3) | 2 (3) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (5)
Insomnia (Psychiatric disorders) | 1 (4) | 1 (1) | 3 (3)
Sleep disorder (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 9 (15) | 3 (3) | 7 (9)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (9) | 2 (2) | 9 (12)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Weight increased (Investigations) | 1 (1) | 0 (0) | 5 (6)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (2) | 5 (8)
Dizziness (Nervous system disorders) | 9 (10) | 5 (5) | 2 (3)
Headache (Nervous system disorders) | 17 (22) | 13 (20) | 11 (14)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Migraine (Nervous system disorders) | 1 (2) | 3 (3) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (2) | 3 (5) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 2 (2) | 2 (3)
Somnolence (Nervous system disorders) | 5 (5) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 3 (4) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 4 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 7 (8) | 7 (8)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4)
Nausea (Gastrointestinal disorders) | 12 (17) | 7 (7) | 6 (6)
Toothache (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (19) | 3 (3) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12) | 5 (5) | 3 (3)
Bone callus excessive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (7) | 8 (9) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (13) | 5 (6) | 9 (13)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 2 (3) | 1 (1) | 6 (6)
Cystitis (Infections and infestations) | 2 (3) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (4) | 3 (3) | 5 (5)
Influenza (Infections and infestations) | 3 (3) | 6 (6) | 3 (3)
Nasopharyngitis (Infections and infestations) | 24 (31) | 18 (26) | 15 (24)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 3 (3) | 3 (4) | 4 (5)
Sinusitis (Infections and infestations) | 7 (8) | 6 (6) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
Two events occured during the trial due to crytals in Dose 2 formulation: hold of all subjects enrolled in Germany (Jun-17) and discontinuation of Dose 2 arm by the sponsor worldwide due to discovery of crystals in the ICH stability batch in Sep-17.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02579759/Prot_SAP_000.pdf